CLINICAL TRIAL: NCT07330011
Title: Inter- and Intra-observer Reliability of the Iowa Level of Assistance (ILoA) Scale for Measuring Postoperative Functional Recovery in Orthopedic Patients: an Observational Study
Brief Title: Inter- and Intra-Observer Reliability of the Iowa Level of Assistance Scale and the Effect of Staff Retraining
Acronym: ILOA
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 522/2025/Oss/IOR
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Joint Replacement; Functional Recovery; Reliability
Keywords: ILOA scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: staff training — A structured training session will be provided to all participating physiotherapists to review the content of the ILoA scale and standardize administration procedures. The training will be delivered by IOR-employed physiotherapists with documented experience in orthopedic patient assessment and in the use of the ILoA scale. For each scale item, potential sources of uncertainty and specific clinical scenarios will be discussed.

SUMMARY:
The aim of this study is to evaluate, in routine clinical practice, the inter- and intra-observer reliability of the Iowa Level of Assistance (ILoA) scale, which is regularly used to assess functional recovery in orthopedic patients. A secondary objective is to investigate the impact of a structured retraining program for healthcare staff on the use of the ILoA scale and to determine whether this intervention influences the reliability indices of the scale.

DETAILED DESCRIPTION:
The study will be conducted among healthcare professionals of the Istituto Ortopedico Rizzoli (IOR). The Iowa Level of Assistance (ILoA) scale has been integrated into the institutional Care Pathways for patients undergoing hip and knee arthroplasty and for patients with femoral fractures, and it is routinely used by rehabilitation healthcare staff.

Retrospective Phase

Pre-training scale assessment To evaluate potential changes in the reliability of the ILoA scale, a retrospective control group will be constructed using video-based assessments that were previously collected as part of a monitoring activity. The procedures for video recording and ILoA scale administration used during this retrospective phase were comparable to those planned for the present study, allowing meaningful comparison of reliability indices.

Prospective Phase

Post-training scale assessment At least three months after completion of the retraining program, a new data collection phase will be conducted. All participating physiotherapists will be asked to independently score the ILoA scale for a group of patients who have undergone hip or knee arthroplasty or osteosynthesis, using standardized video recordings. Assessments will be performed anonymously by the observers.

To evaluate intra-observer reliability, the scoring procedure will be repeated on two separate occasions at least two weeks apart, using the same video recordings.

ELIGIBILITY:
Inclusion Criteria:

* For Observers (Physiotherapists):

All physiotherapists working at the main Istituto Ortopedico Rizzoli (IOR) site in Bologna or at the two satellite sites in Argenta and Bagheria.

Physiotherapists must have the role of observers in the study. All physiotherapists affiliated with the SAITeR service who have previously received initial training in the use of the ILoA scale; newly hired staff must have completed the specific training pathway.

For Patients:

Patients admitted to IOR Bologna or Argenta for whom administration of the ILoA scale is part of routine clinical practice.

Patients undergoing primary hip or knee arthroplasty for osteoarthritis. Patients undergoing revision hip or knee arthroplasty. Patients undergoing hip arthroplasty or osteosynthesis for femoral fracture.

Exclusion Criteria:

* Refusal or inability to provide informed consent (for both physiotherapists and patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit both patients and physiotherapists. Patients will be those who, according to routine clinical practice, are assessed using the Iowa Level of Assistance (ILoA) scale and who provide informed consent to participate in the study and to be video-recorded. Physiotherapists will administer the ILoA scale during clinical assessments and, subsequently, will reassess patient performance by reviewing the video recordings of the participating patients.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Inter- and Intra-Observer Reliability of the Iowa Level of Assistance (ILoA) Scale | Baseline (pre-training) and within 6 months after completion of staff training.
  The Iowa Level of Assistance (ILoA) scale assesses five functional activities: moving to a sitting position, static standing, walking, stair negotiation, and gait speed. For each activity, a score is assigned based on the level of assistance provided, ranging from 0 (independent) to 6 (activity not performed), and on the type of assistive device used, ranging from 0 (no device) to 5 (use of a walker). The total ILoA score ranges from 0 (minimal assistance) to 50 (maximal assistance).
  The primary outcome of this study is the inter- and intra-observer reliability of the ILoA scale. Inter-observer reliability will be defined as the level of agreement between different observers assessing the same patient under identical clinical conditions, while intra-observer reliability will be defined as the level of agreement between repeated assessments performed by the same observer on the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Morri, Principal Investigator — IRCCS Istotuto Ortopedico Rizzoli
Locations (1):
- SAITeR IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Yang Y, Wang Y, Zhou Y, Chen C, Xing D. Reliability of functional gait assessment in patients with Parkinson disease: Interrater and intrarater reliability and internal consistency. Medicine (Baltimore). 2016 Aug;95(34):e4545. doi: 10.1097/MD.0000000000004545. PMID 27559954
- [Result] Shields RK, Enloe LJ, Evans RE, Smith KB, Steckel SD. Reliability, validity, and responsiveness of functional tests in patients with total joint replacement. Phys Ther. 1995 Mar;75(3):169-76; discussion 176-9. doi: 10.1093/ptj/75.3.169. PMID 7870749
- [Result] Morri M, Franchini N, Gerini G, Morabito R, Pignotti E, Benedetti MG, Marchese O, Zanotti E. Measuring functional performance at discharge from hospital after total joint arthroplasty as a pre-requisite for planning early rehabilitation: a prognostic study. Orthop Nurs. 2015 Mar-Apr;34(2):95-100. doi: 10.1097/NOR.0000000000000126. PMID 25785619
- [Result] Benedetti MG, Franchignoni F, Morri M, Franchini N, Natali E, Giordano A. Rasch analysis of the Iowa Level of Assistance Scale in patients with total hip and knee arthroplasty. Int J Rehabil Res. 2014 Jun;37(2):118-24. doi: 10.1097/MRR.0000000000000043. PMID 24406302